CLINICAL TRIAL: NCT00085943
Title: See Detailed Description
Brief Title: KALETRA Or LEXIVA With Ritonavir Combined With EPIVIR And Abacavir In Naive Subjects Over 48 Weeks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Cheri Hudson; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100732
Record Dates: First submitted 2004-06-17; First posted 2004-06-21 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: HIV Infection; Infection, Human Immunodeficiency Virus
Keywords: ritonavir; abacavir; HIV; lopinavir; lamivudine; fosamprenavir; Epzicom
MeSH Terms: conditions — HIV Infections; Infections; Acquired Immunodeficiency Syndrome | interventions — fosamprenavir; Ritonavir; lopinavir-ritonavir drug combination; Lamivudine; abacavir; abacavir, lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: LEXIVA (GW433908)
Drug: Ritonavir
Drug: KALETRA
Drug: EPIVIR
Drug: Ziagen
Drug: Abacavir/Lamivudine
Drug: Fosamprenavir
  Other Names: LEXIVA (GW433908); Ritonavir; Ziagen; KALETRA; Abacavir/Lamivudine; EPIVIR

SUMMARY:
This study will compare the ability of fosamprenavir 700 mg with ritonavir 100 mg twice a day or lopinavir 400 mg with ritonavir 100 mg twice a day both combined with a fixed dose combination tablet of abacavir 600 mg and lamivudine 300 mg once a day to suppress virus levels of HIV to less than 400 copies/mL of blood. In addition we will study the safety and tolerability of these compounds over the 48 week study period in patients naive to anti-HIV therapy.

DETAILED DESCRIPTION:
A Phase IIIB, Randomized, Open-Label, Multicenter Study of the Safety and Efficacy of GW433908 (700mg BID) plus ritonavir (100mg BID) Versus Lopinavir/ritonavir (400mg/100mg BID) when Administered in Combination with the Abacavir/Lamivudine (600mg/300mg) Fixed-Dose Combination Tablet QD in Antiretroviral-Naive HIV-1 Infected Adults Over 48 Weeks

ELIGIBILITY:
Inclusion Criteria:

* HIV infected subjects that are naive to anti-HIV therapy.
* History of a positive HIV test.
* At least 1000 copies/mL of HIV in their blood as screening.

Exclusion Criteria:

* Active HIV-related diseases.
* Taking other investigational drugs.
* Pregnant or breastfeeding females.
* Not be suitable to participate per investigator opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 866
Dates: Start 2004-05

PRIMARY OUTCOMES:
Proportion of subjects with plasma HIV-1 RNA <400 copies/mL at Week 48. Proportion of subjects who permanently discontinue randomized treatment due to adverse events.

SECONDARY OUTCOMES:
Proportion of subjects with plasma HIV-1 RNA <400 copies/mL at Week 48. Proportion of subjects who permanently discontinue randomized treatment due to adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Pharm.D., Study Director — GlaxoSmithKline
Locations (92):
- United States (45):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Lynchburg, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
- GSK Investigational Site, Vienna, Austria
- Belgium (5):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Charleroi
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (5):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Denis
- Germany (6):
  - GSK Investigational Site, Fürth, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- Italy (6):
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Busto Arsizio (VA), Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
- GSK Investigational Site, Riga, Latvia
- GSK Investigational Site, Luxembourg, Luxembourg
- Poland (3):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Wroclaw
- GSK Investigational Site, Cascais, Portugal
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași
- Spain (9):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Tarrasa, Barcelona
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo ( Pontevedra)
- Switzerland (3):
  - GSK Investigational Site, Lugano
  - GSK Investigational Site, Olten
  - GSK Investigational Site, Sankt Gallen

REFERENCES:
- [Background] Eron J Jr, Yeni P, Gathe J Jr, Estrada V, DeJesus E, Staszewski S, Lackey P, Katlama C, Young B, Yau L, Sutherland-Phillips D, Wannamaker P, Vavro C, Patel L, Yeo J, Shaefer M; KLEAN study team. The KLEAN study of fosamprenavir-ritonavir versus lopinavir-ritonavir, each in combination with abacavir-lamivudine, for initial treatment of HIV infection over 48 weeks: a randomised non-inferiority trial. Lancet. 2006 Aug 5;368(9534):476-82. doi: 10.1016/S0140-6736(06)69155-1. PMID 16890834